CLINICAL TRIAL: NCT05392816
Title: Non-heme Iron Absorption From Single Meals of Fava Bean Protein, Beef Protein and Cod Protein in Healthy Females in Fertile Ages
Brief Title: Non-heme Iron Absorption From Single Meals of Fava Bean Protein, Beef Protein and Cod Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 573-18
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Healthy; Nutrition, Healthy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Meals are served from identical plastic boxes. Participants are served the meals in a separate room from preparation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group 1. Texturized fava protein meal and beef protein meal (Other): Participants recruited to study group 1 will be served a meal with fava bean protein (B) and beef protein (A), each meal twice which in total brings four meals on four consecutive days as fasting breakfast. Meals are served in the order BBAA
  Interventions: Other: Single meal non-heme iron absorption
- Study group 2. Texturized fava protein meal and cod protein meal (Other): Participants recruited to study group 1 will be served a meal with fava bean protein (B) and cod protein (A), each meal twice which in total brings four meals on four consecutive days as fasting breakfast. Meals are served in the order BBAA
  Interventions: Other: Single meal non-heme iron absorption

INTERVENTIONS:
Other: Single meal non-heme iron absorption — Two study groups, each designed as cross-over single-blinded iron isotope trials in apparent healthy Swedish women of the ages 18-45 years. Each participant serves as their own control. Meals are tagged with radiolabeled non-heme iron 55Fe and 59Fe.

SUMMARY:
The aim of this study is to investigate the non-heme iron absorption from single meals of texturized fava bean protein, which has been suggested as a protein source suitable for replacement of meat, compared to the non-heme iron absorption from beef protein and cod protein meals. The study participants are women of fertile ages, which is one of the main groups at risk of developing iron deficiency. Since a dietary shift towards increasingly plant based is being pushed, investigating nutritional effects of such a shift is essential to avoid potential negative effects such as an increase of nutritional deficiencies. The study includes two cross-over single-blinded iron isotope trials in apparent healthy Swedish women of the ages 18-45 years, each of whom served as their own control. Participants will be served matched test meals containing beef and fava bean protein (Study 1), or cod and fava bean protein (Study 2) with radiolabeled non-heme iron 55Fe and 59Fe. Absorption of non-heme iron from test meals will be measured by whole-body counting, and erythrocyte incorporation by liquid scintillation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-45
* Is tolerant to intake of fava bean
* Eats fish and meat
* Feels healthy
* Can eat a breakfast consisting of three potato-based patties

Exclusion Criteria:

* Other sex than female
* Age <18 and >45
* Has an ongoing infection
* Is vegetarian
* Is pregnant or lactating
* Takes iron supplements

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
59Fe non-heme iron absorption from cod and beef protein meals | 5 weeks
  Absorption of 59Fe, which is added to the animal protein meals, will be measured by a whole body counter which enables measurement of absolute value.
55Fe non-heme iron absorption from fava bean protein meals. | 5 weeks
  The absorption quota of 59Fe/55Fe is measured by erythrocyte incorporation, analyzed by liquid scintillation. The absorbance quota, in combination with the absolute value of the whole body counter, will be used to calculate the absorbance of 55Fe which is added to the fava bean meals

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Sofie Sandberg, Professor, Principal Investigator — Chalmers University of Technology
Locations (1):
- Chalmers University of Technology, Division of Food Science, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided